CLINICAL TRIAL: NCT05051579
Title: A Phase 2 Study of Once-Daily LY3502970 Compared With Placebo in Participants Who Have Obesity or Are Overweight With Weight-Related Comorbidities
Brief Title: A Study of LY3502970 in Participants With Obesity or Overweight With Weight-related Comorbidities
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18210; J2A-MC-GZGI (Other: Eli Lilly and Company); 2021-002805-88 (EudraCT Number)
Record Dates: First submitted 2021-09-17; First posted 2021-09-21 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Obesity; Overweight and Obesity
MeSH Terms: conditions — Obesity; Overweight | interventions — orforglipron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- 12 milligram (mg) LY3502970 (Experimental): Participants received maintenance dose 12 mg with dose escalation starting from 3 mg,6 mg and then 12 mg LY3502970 administered orally once daily until 36 weeks.
  Interventions: Drug: LY3502970
- 24 mg LY3502970 (Experimental): Participants received maintenance dose 24 mg with dose escalation starting from 3 mg, 6 mg, 8 mg,12 mg and then 24 mg LY3502970 administered orally once daily until 36 weeks.
  Interventions: Drug: LY3502970
- 36 mg-1 LY3502970 (Experimental): Participants received maintenance dose 36 mg with dose escalation starting from 2 mg, 3 mg, 6 mg, 8 mg, 12 mg, 24 mg and then 36 mg LY3502970 administered orally once daily until 36 weeks.
  Interventions: Drug: LY3502970
- 36 mg-2 LY3502970 (Experimental): Participants received maintenance dose 36 mg with dose escalation starting from 3 mg, 6 mg,12 mg, 24 mg and then 36 mg LY3502970 administered orally once daily until 36 weeks.
  Interventions: Drug: LY3502970
- 45 mg-1 LY3502970 (Experimental): Participants received maintenance dose 45 mg with dose escalation starting from 3 mg, 6 mg, 8 mg, 12 mg, 24 mg, 36 mg and then 45 mg LY3502970 administered orally once daily until 36 weeks.
  Interventions: Drug: LY3502970
- 45 mg-2 LY3502970 (Experimental): Participants received maintenance dose 45 mg with dose escalation starting from 2 mg, 3 mg, 6 mg, 12 mg, 24 mg, 36 mg and then 45 mg LY3502970 administered orally once daily until 36 weeks.
  Interventions: Drug: LY3502970
- Placebo (Placebo Comparator): Participants received placebo administered orally once daily until 36 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3502970 — Administered orally
  Arms: 12 milligram (mg) LY3502970; 24 mg LY3502970; 36 mg-1 LY3502970; 36 mg-2 LY3502970; 45 mg-1 LY3502970; 45 mg-2 LY3502970
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of the study was to assess the effect of LY3502970 in participants who have obesity or are overweight.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) of ≥30-kilogram square meter (kg/m²)
* Have a BMI ≥27 kg/m² and <30 kg/m² with at least 1 of the following weight-related comorbidities eg; [Have hypertension, or dyslipidemia, cardiovascular disease]
* Have had a stable body weight for the 3 months prior to randomization (not more than 5% body weight gain and/or loss)

Exclusion Criteria:

* Have any prior diagnosis of diabetes
* Have a prior or planned surgical treatment for obesity
* Have obesity induced by other endocrinological disorders or diagnosed monogenetic or syndromic forms of obesity
* Have renal impairment measured as estimated glomerular filtration rate (eGFR) <30 milliliter (mL)/minute (min)/1.73 m²
* Have a history of acute chronic pancreatitis
* Have a history of significant active or unstable Major Depressive Disorder (MDD) or other severe psychiatric disorder (for example, schizophrenia, bipolar disorder, or other serious mood or anxiety disorder) within the last 2 years Note: Participants with MDD or generalized anxiety disorder whose disease state is considered stable for the past 2 years and expected to remain stable throughout the course of the study, may be considered for inclusion if they are not on excluded medications.

Within 3 months prior to screening:

* Have poorly controlled hypertension
* Have history of acute myocardial infarction
* Have history of cerebrovascular accident (stroke)
* Had hospitalization due to congestive heart failure (CHF)
* Have cancer
* Have human immunodeficiency virus (HIV) and/or positive HIV antibodies historically or at screening
* Have hepatitis B and/or positive hepatitis B surface antigen

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-5615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (35):
- United States (18):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - John Muir Physician Network Research Center, Concord, California
  - NorCal Medical Research, Inc, Greenbrae, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Norcal Endocrinology & Internal Medicine, San Ramon, California
  - Elite Clinical Trials, Blackfoot, Idaho
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Premier Research, Trenton, New Jersey
  - Lillestol Research, Fargo, North Dakota
  - Intend Research, LLC, Norman, Oklahoma
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Preferred Primary Care Physicians, Preferred Clinical Research-St. Clair, Pittsburgh, Pennsylvania
  - Dallas Diabetes Research Center, Dallas, Texas
  - Diabetes and Thyroid Center of Fort Worth, Fort Worth, Texas
  - Texas Diabetes & Endocrinology, P.A., Round Rock, Texas
  - National Clinical Research, Inc, Richmond, Virginia
  - St. Vincent Hospital d/b/a Prevea Health, Green Bay, Wisconsin
- Canada (6):
  - C-health Research, Calgary, Alberta
  - Wharton Medical Clinic, Hamilton, Ontario
  - Bluewater Clinical Research Group Inc., Sarnia, Ontario
  - Centre Médical et Professionnel de l'Ouest de Portneuf, Saint-Marc-des-Carrieres, Quebec
  - Alpha Recherche Clinique, Québec
  - ALPHA Recherche Clinique, Québec
- Hungary (9):
  - Studium Egeszseghaz Kft, Kalocsa, Bács-Kiskun county
  - Bugát Pál Kórház, Gyöngyös, Heves County
  - DRC Gyógyszervizsgáló Központ, Balatonfüred, Veszprém megye
  - Kanizsai Dorottya Korhaz, Nagykanizsa, Zala County
  - Szent Margit Rendelőintézet Nonprofit Kft, Budapest
  - Clinexpert Kft., Budapest
  - TRANTOR'99 Bt. Anyagcsere Centrum, Budapest
  - Strazsahegy Medicina Bt., Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
- Puerto Rico (2):
  - Puerto Rico Medical Research, Ponce
  - Research and Cardiovascular Corp., Ponce

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Wharton S, Rosenstock J, Konige M, Lin Y, Duffin K, Wilson J, Banerjee H, Pirro V, Kazda C, Mather K. Treatment with orforglipron, an oral glucagon like peptide-1 receptor agonist, is associated with improvements of CV risk biomarkers in participants with type 2 diabetes or obesity without diabetes. Cardiovasc Diabetol. 2025 Jun 6;24(1):240. doi: 10.1186/s12933-025-02781-x. PMID 40481478
- [Derived] Wharton S, Blevins T, Connery L, Rosenstock J, Raha S, Liu R, Ma X, Mather KJ, Haupt A, Robins D, Pratt E, Kazda C, Konig M; GZGI Investigators. Daily Oral GLP-1 Receptor Agonist Orforglipron for Adults with Obesity. N Engl J Med. 2023 Sep 7;389(10):877-888. doi: 10.1056/NEJMoa2302392. Epub 2023 Jun 23. PMID 37351564
- See also: A Study of LY3502970 in Participants With Obesity or Overweight With Weight-related Comorbidities — https://trials.lillytrialguide.com/en-US/trial/1R7BP1Yw5t6roV3ZWFGzYQ

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For maintenance doses of LY3502970: 12, 24, 36, and 45 milligram (mg), the initial dose will be 2 or 3 mg followed by additional escalation steps as appropriate. The dose-escalation varied by dose group where the target maintenance dose was achieved between Weeks 5 and 16.
Groups:
- 12 mg LY3502970: Participants received maintenance dose 12 mg with dose escalation starting from 3 mg, 6 mg and then 12 mg LY3502970 administered orally once daily until 36 weeks.
- 36 mg -1 LY3502970: Participants received maintenance dose 36 mg with dose escalation starting from 2 mg, 3 mg, 6 mg, 8 mg, 12 mg, 24 mg and then 36 mg LY3502970 administered orally once daily until 36 weeks.
- 36 mg -2 LY3502970: Participants received maintenance dose 36 mg with dose escalation starting from 3 mg, 6 mg,12 mg, 24 mg and then 36 mg LY3502970 administered orally once daily until 36 weeks.
- 45 mg -1 LY3502970: Participants received maintenance dose 45 mg with dose escalation starting from 3 mg, 6 mg, 8 mg, 12 mg, 24 mg, 36 mg and then 45 mg LY3502970 administered orally once daily until 36 weeks.
- 45 mg -2 LY3502970: Participants received maintenance dose 45 mg with dose escalation starting from 2 mg, 3 mg, 6 mg, 12 mg, 24 mg, 36 mg and then 45 mg LY3502970 administered orally once daily until 36 weeks.
Period: Overall Study
Arm/Group | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg -1 LY3502970 | 36 mg -2 LY3502970 | 45 mg -1 LY3502970 | 45 mg -2 LY3502970 | Placebo
Started | 50 | 53 | 29 | 29 | 31 | 30 | 50
Completed | 44 | 46 | 27 | 24 | 23 | 28 | 43
Not Completed | 6 | 7 | 2 | 5 | 8 | 2 | 7
Not completed — Withdrawal by Subject | 3 | 5 | 2 | 1 | 4 | 0 | 4
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Subject Unable to Visit Due to Working Out of Town | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 2 | 1 | 0 | 4 | 1 | 2 | 0
Not completed — Inadvertent Enrollment | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Subject Could not Tolerate Investigational Product (IP) and was Taken Off | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Patient was Initially Long Term Follow-up But Contacted and came to Site After Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 12 mg LY3502970: Participants received maintenance dose 12 mg with dose escalation starting from 3 mg,6 mg and then 12 mg LY3502970 administered orally once daily until 36 weeks.
- Total: Total of all reporting groups
Arm/Group | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg -1 LY3502970 | 36 mg -2 LY3502970 | 45 mg -1 LY3502970 | 45 mg -2 LY3502970 | Placebo | Total
Number analyzed (Participants) | 50 | 53 | 29 | 29 | 31 | 30 | 50 | 272
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.80 (10.51) | 57.00 (9.09) | 56.30 (11.83) | 55.40 (10.93) | 56.50 (10.74) | 50.90 (12.58) | 54.00 (8.82) | 54.20 (10.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 18 | 18 | 19 | 16 | 29 | 161
  Male | 19 | 23 | 11 | 11 | 12 | 14 | 21 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 6 | 4 | 2 | 4 | 7 | 5 | 39
  Not Hispanic or Latino | 38 | 46 | 23 | 26 | 25 | 22 | 43 | 223
  Unknown or Not Reported | 1 | 1 | 2 | 1 | 2 | 1 | 2 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 6 | 4 | 4 | 1 | 0 | 1 | 19
  White | 47 | 46 | 25 | 25 | 29 | 30 | 45 | 247
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 9 | 11 | 5 | 3 | 9 | 5 | 6 | 48
  Hungary | 6 | 5 | 3 | 6 | 3 | 3 | 5 | 31
  United States | 35 | 37 | 21 | 20 | 19 | 22 | 39 | 193
Baseline Body Weight [Mean (Standard Deviation); unit: Kilograms (kg)] | 107.49 (25.34) | 112.05 (30.18) | 107.78 (22.45) | 108.84 (28.52) | 105.23 (20.40) | 110.85 (28.11) | 107.57 (25.24) | 108.68 (26.03)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Body Weight in LY3502970 and Placebo
Description: Least Squares (LS) mean was determined by mixed model repeated measures (MMRM) model with Baseline + Baseline BMI Group + Sex + Treatment + Time + Treatment*Time (Type III sum of squares) as variables. Variance-Covariance structure (Actual Value) = Unstructured. Variance-Covariance structure (Percent Change from Baseline) = Unstructured.
Time Frame: Baseline, Week 26
Population: All randomized participants who received at least one dose of study drug and had baseline and at least one post-baseline body weight value.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Groups:
- 36 mg LY3502970: Participants received maintenance dose 36 mg with dose escalation starting from 2 mg, 3 mg, 6 mg, 8 mg, 12 mg, 24 mg and then 36 mg LY3502970 in LY 36mg-1 and dose escalation starting from 3 mg, 6 mg,12 mg, 24 mg and then 36 mg LY3502970 in LY 36mg-2 administered orally once daily until 36 weeks.
- 45 mg LY3502970: Participants received maintenance dose 45 mg with dose escalation starting from 3 mg, 6 mg, 8 mg, 12 mg, 24 mg, 36 mg and then 45 mg LY3502970 in LY 45mg-1 and dose escalation starting from 2 mg, 3 mg, 6 mg, 12 mg, 24 mg, 36 mg and then 45 mg LY3502970 in LY 45mg-2 administered orally once daily until 36 weeks.
Arm/Group | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg LY3502970 | 45 mg LY3502970 | Placebo
Number analyzed (Participants) | 44 | 51 | 56 | 57 | 48
Percent change | -8.6 (0.85) | -11.2 (0.82) | -12.3 (0.77) | -12.6 (0.75) | -2.0 (0.81)
Statistical Analysis 1: Comparison: 12 mg LY3502970 vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -6.5, 95% CI 2-sided [-8.9 to -4.2]
Statistical Analysis 2: Comparison: 24 mg LY3502970 vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -9.2, 95% CI 2-sided [-11.5 to -6.9]
Statistical Analysis 3: Comparison: 36 mg LY3502970 vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -10.2, 95% CI 2-sided [-12.4 to -8.0]
Statistical Analysis 4: Comparison: 45 mg LY3502970 vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -10.6, 95% CI 2-sided [-12.7 to -8.4]

2. Secondary Outcome: Percent Change From Baseline in Body Weight in LY3502970 and Placebo
Description: LS mean was determined by MMRM model with Baseline + Baseline BMI Group + Sex + Treatment + Time + Treatment*Time (Type III sum of squares) as variables. Variance-Covariance structure (Actual Value) = Unstructured. Variance-Covariance structure (Percent Change from Baseline) = Unstructured.
Time Frame: Baseline, Week 36
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg LY3502970 | 45 mg LY3502970 | Placebo
Number analyzed (Participants) | 44 | 51 | 56 | 57 | 48
Percent change | -9.4 (1.05) | -12.5 (1.01) | -13.5 (0.95) | -14.7 (0.94) | -2.3 (1.00)
Statistical Analysis 1: Comparison: 12 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -7.1, 95% CI 2-sided [-9.9 to -4.2]
Statistical Analysis 2: Comparison: 24 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -10.1, 95% CI 2-sided [-12.9 to -7.3]
Statistical Analysis 3: Comparison: 36 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -11.1, 95% CI 2-sided [-13.8 to -8.4]
Statistical Analysis 4: Comparison: 45 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -12.3, 95% CI 2-sided [-15.0 to -9.6]

3. Secondary Outcome: Change From Baseline in Body Weight in LY3502970 and Placebo
Description: as for outcome 2
Time Frame: Baseline, Week 26
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg LY3502970 | 45 mg LY3502970 | Placebo
Number analyzed (Participants) | 44 | 51 | 56 | 57 | 48
kg | -9.0 (0.90) | -12.3 (0.86) | -12.9 (0.82) | -13.3 (0.79) | -2.1 (0.86)
Statistical Analysis 1: Comparison: 12 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -6.9, 95% CI 2-sided [-9.3 to -4.4]
Statistical Analysis 2: Comparison: 24 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -10.2, 95% CI 2-sided [-12.5 to -7.8]
Statistical Analysis 3: Comparison: 36 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -10.8, 95% CI 2-sided [-13.1 to -8.5]
Statistical Analysis 4: Comparison: 45 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -11.2, 95% CI 2-sided [-13.5 to -8.9]

4. Secondary Outcome: Change From Baseline in Body Weight in LY3502970 and Placebo
Description: as for outcome 2
Time Frame: Baseline, Week 36
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg LY3502970 | 45 mg LY3502970 | Placebo
Number analyzed (Participants) | 44 | 51 | 56 | 57 | 48
kg | -9.8 (1.10) | -13.6 (1.06) | -14.2 (1.00) | -15.4 (0.98) | -2.4 (1.05)
Statistical Analysis 1: Comparison: 12 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -7.4, 95% CI 2-sided [-10.4 to -4.3]
Statistical Analysis 2: Comparison: 24 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -11.2, 95% CI 2-sided [-14.2 to -8.3]
Statistical Analysis 3: Comparison: 36 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -11.8, 95% CI 2-sided [-14.7 to -9.0]
Statistical Analysis 4: Comparison: 45 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -13.0, 95% CI 2-sided [-15.8 to -10.2]

5. Secondary Outcome: Change From Baseline in Waist Circumference in LY3502970 and Placebo
Description: as for outcome 2
Time Frame: Baseline, Week 26
Population: All randomized participants who received at least one dose of study drug and had baseline and at least one post-baseline body waist circumference value.
Measure: Least Squares Mean (Standard Error); unit: centimeter (cm)
Arm/Group | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg LY3502970 | 45 mg LY3502970 | Placebo
Number analyzed (Participants) | 43 | 49 | 52 | 57 | 48
centimeter (cm) | -8.0 (1.03) | -8.8 (1.00) | -10.1 (0.94) | -12.2 (0.93) | -3.6 (0.99)
Statistical Analysis 1: Comparison: 12 mg LY3502970 vs Placebo; Test type: Other; p = 0.002, Mixed Models Analysis; LS Mean difference (Final Values) = -4.4, 95% CI 2-sided [-7.2 to -1.6]
Statistical Analysis 2: Comparison: 24 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -5.2, 95% CI 2-sided [-8.0 to -2.4]
Statistical Analysis 3: Comparison: 36 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -6.5, 95% CI 2-sided [-9.2 to -3.8]
Statistical Analysis 4: Comparison: 45 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -8.7, 95% CI 2-sided [-11.3 to -6.0]

6. Secondary Outcome: Change From Baseline in Waist Circumference in LY3502970 and Placebo
Description: as for outcome 2
Time Frame: Baseline, Week 36
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg LY3502970 | 45 mg LY3502970 | Placebo
Number analyzed (Participants) | 43 | 49 | 52 | 57 | 48
cm | -9.6 (1.18) | -11.2 (1.15) | -10.6 (1.06) | -13.6 (1.07) | -4.0 (1.12)
Statistical Analysis 1: Comparison: 12 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -5.6, 95% CI 2-sided [-8.8 to -2.4]
Statistical Analysis 2: Comparison: 24 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -7.2, 95% CI 2-sided [-10.3 to -4.0]
Statistical Analysis 3: Comparison: 36 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -6.6, 95% CI 2-sided [-9.7 to -3.6]
Statistical Analysis 4: Comparison: 45 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -9.6, 95% CI 2-sided [-12.7 to -6.6]

7. Secondary Outcome: Change From Baseline in BMI in LY3502970 and Placebo
Description: as for outcome 2
Time Frame: Baseline, Week 26
Population: All randomized participants who received at least one dose of study drug and had baseline and at least one post-baseline BMI value.
Measure: Least Squares Mean (Standard Error); unit: kilograms per meter square (kg/m^2)
Arm/Group | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg LY3502970 | 45 mg LY3502970 | Placebo
Number analyzed (Participants) | 44 | 51 | 56 | 57 | 48
kilograms per meter square (kg/m^2) | -3.2 (0.31) | -4.2 (0.30) | -4.6 (0.28) | -4.7 (0.27) | -0.8 (0.29)
Statistical Analysis 1: Comparison: 12 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -2.4, 95% CI 2-sided [-3.2 to -1.6]
Statistical Analysis 2: Comparison: 24 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -3.5, 95% CI 2-sided [-4.3 to -2.6]
Statistical Analysis 3: Comparison: 36 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -3.8, 95% CI 2-sided [-4.6 to 3.0]
Statistical Analysis 4: Comparison: 45 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -3.9, 95% CI 2-sided [-4.7 to -3.1]

8. Secondary Outcome: Change From Baseline in BMI in LY3502970 and Placebo
Description: as for outcome 2
Time Frame: Baseline, Week 36
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg LY3502970 | 45 mg LY3502970 | Placebo
Number analyzed (Participants) | 44 | 51 | 56 | 57 | 48
kg/m^2 | -3.4 (0.38) | -4.7 (0.36) | -5.0 (0.34) | -5.5 (0.34) | -0.9 (0.36)
Statistical Analysis 1: Comparison: 12 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -2.5, 95% CI 2-sided [-3.6 to -1.5]
Statistical Analysis 2: Comparison: 24 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -3.8, 95% CI 2-sided [-4.8 to -2.8]
Statistical Analysis 3: Comparison: 36 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -4.2, 95% CI 2-sided [-5.2 to -3.2]
Statistical Analysis 4: Comparison: 45 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -4.6, 95% CI 2-sided [-5.6 to -3.6]

9. Secondary Outcome: Percentage of Participants With >=5% Body Weight Loss
Description: Percentage of participants with >=5% body weight loss was reported.
Time Frame: Week 26
Population: All randomized participants who received at least one dose of study drug and had baseline and at least one post-baseline value for ≥5% body weight reduction.
Measure: Number; unit: percentage of participants
Arm/Group | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg LY3502970 | 45 mg LY3502970 | Placebo
Number analyzed (Participants) | 44 | 51 | 56 | 57 | 48
percentage of participants | 74.39 | 88.84 | 89.46 | 87.26 | 22.88
Statistical Analysis 1: Comparison: 12 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 9.96, 95% CI 2-sided [3.61 to 27.44]
Statistical Analysis 2: Comparison: 24 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 27.97, 95% CI 2-sided [8.15 to 96.01]
Statistical Analysis 3: Comparison: 36 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 27.36, 95% CI 2-sided [8.71 to 85.91]
Statistical Analysis 4: Comparison: 45 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 23.59, 95% CI 2-sided [7.65 to 72.77]

10. Secondary Outcome: Percentage of Participants With >=10% Body Weight Loss
Description: Percentage of participants with >=10% body weight loss was reported.
Time Frame: Week 26
Population: All randomized participants who received at least one dose of study drug and had baseline and at least one post-baseline value for ≥10% body weight reduction.
Measure: Number; unit: percentage of participants
Arm/Group | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg LY3502970 | 45 mg LY3502970 | Placebo
Number analyzed (Participants) | 44 | 51 | 56 | 57 | 48
percentage of participants | 39.39 | 56.61 | 71.30 | 69.86 | 2.25
Statistical Analysis 1: Comparison: 12 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 19.93, 95% CI 2-sided [3.47 to 114.40]
Statistical Analysis 2: Comparison: 24 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 39.52, 95% CI 2-sided [6.95 to 224.83]
Statistical Analysis 3: Comparison: 36 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 74.97, 95% CI 2-sided [13.16 to 427.18]
Statistical Analysis 4: Comparison: 45 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 72.23, 95% CI 2-sided [12.62 to 413.21]

11. Secondary Outcome: Percentage of Participants With >=5% Body Weight Loss
Description: Percentage of participants with >=5% body weight loss was reported.
Time Frame: Week 36
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg LY3502970 | 45 mg LY3502970 | Placebo
Number analyzed (Participants) | 44 | 51 | 56 | 57 | 48
percentage of participants | 72.00 | 89.47 | 92.05 | 90.44 | 24.02
Statistical Analysis 1: Comparison: 12 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 7.79, 95% CI 2-sided [2.90 to 20.92]
Statistical Analysis 2: Comparison: 24 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 25.07, 95% CI 2-sided [7.49 to 83.91]
Statistical Analysis 3: Comparison: 36 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 34.76, 95% CI 2-sided [8.17 to 147.86]
Statistical Analysis 4: Comparison: 45 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 28.01, 95% CI 2-sided [8.15 to 96.29]

12. Secondary Outcome: Percentage of Participants With >=10% Body Weight Loss
Description: Percentage of participants with >=10% body weight loss was reported.
Time Frame: Week 36
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | 12 mg LY3502970 | 24 mg LY3502970 | 36 mg LY3502970 | 45 mg LY3502970 | Placebo
Number analyzed (Participants) | 44 | 51 | 56 | 57 | 48
percentage of participants | 46.50 | 61.88 | 74.75 | 69.07 | 8.85
Statistical Analysis 1: Comparison: 12 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 8.27, 95% CI 2-sided [2.59 to 26.45]
Statistical Analysis 2: Comparison: 24 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 15.64, 95% CI 2-sided [4.83 to 50.68]
Statistical Analysis 3: Comparison: 36 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 27.24, 95% CI 2-sided [8.39 to 88.38]
Statistical Analysis 4: Comparison: 45 mg LY3502970 vs Placebo; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 20.88, 95% CI 2-sided [6.59 to 66.17]

ADVERSE EVENTS:
Time Frame: Baseline through Week 38 (36 weeks with 2 weeks safety follow up)
Description: All randomized participants who received at least one dose of study drug regardless of adherence to study drug. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | 12 mg LY3502970 | 24 mg LY3502970 | 36 Mg-1 LY3502970 | 36 Mg-2 LY3502970 | 45 Mg-1 LY3502970 | 45 Mg-2 LY3502970 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/53 | 0/29 | 0/29 | 0/31 | 0/30 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 2/53 | 0/29 | 3/29 | 2/31 | 0/30 | 0/50
Other Adverse Events (participants affected / at risk) | 35/50 | 46/53 | 23/29 | 25/29 | 26/31 | 24/30 | 27/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 12 mg LY3502970 (N=50) | 24 mg LY3502970 (N=53) | 36 Mg-1 LY3502970 (N=29) | 36 Mg-2 LY3502970 (N=29) | 45 Mg-1 LY3502970 (N=31) | 45 Mg-2 LY3502970 (N=30) | Placebo (N=50)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal vein thrombosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitreoretinal traction syndrome (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 12 mg LY3502970 (N=50) | 24 mg LY3502970 (N=53) | 36 Mg-1 LY3502970 (N=29) | 36 Mg-2 LY3502970 (N=29) | 45 Mg-1 LY3502970 (N=31) | 45 Mg-2 LY3502970 (N=30) | Placebo (N=50)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 4 (5) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 4 (5) | 0 (0) | 2 (2) | 2 (2) | 1 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 12 (16) | 17 (21) | 8 (8) | 7 (10) | 6 (8) | 4 (5) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 12 (23) | 19 (29) | 1 (1) | 4 (5) | 5 (5) | 10 (16) | 5 (6)
Dyspepsia (Gastrointestinal disorders) | 8 (11) | 4 (4) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 3 (4)
Eructation (Gastrointestinal disorders) | 9 (15) | 11 (14) | 5 (5) | 2 (2) | 2 (2) | 6 (9) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 5 (6) | 3 (3) | 4 (5) | 4 (6) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 25 (39) | 31 (50) | 12 (18) | 14 (18) | 13 (28) | 11 (23) | 5 (6)
Vomiting (Gastrointestinal disorders) | 13 (23) | 17 (33) | 8 (11) | 4 (9) | 9 (14) | 8 (15) | 3 (3)
Chills (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 7 (8) | 4 (4) | 2 (2) | 4 (5) | 4 (6) | 1 (1)
Covid-19 (Infections and infestations) | 9 (11) | 9 (9) | 4 (4) | 7 (7) | 5 (5) | 5 (5) | 9 (9)
Nasopharyngitis (Infections and infestations) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (4) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 4 (5) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 5 (5) | 2 (3) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 8 (11) | 3 (3) | 2 (2) | 4 (6) | 2 (3) | 5 (7)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0/19 (0) | 0/23 (0) | 1/11 (1) | 0/11 (0) | 0/12 (0) | 0/14 (0) | 0/21 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1/19 (1) | 0/23 (0) | 0/11 (0) | 0/11 (0) | 0/12 (0) | 0/14 (0) | 0/21 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0/31 (0) | 0/30 (0) | 0/18 (0) | 1/18 (1) | 1/19 (1) | 0/16 (0) | 0/29 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0/31 (0) | 0/30 (0) | 1/18 (1) | 0/18 (0) | 0/19 (0) | 0/16 (0) | 0/29 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT05051579/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT05051579/SAP_001.pdf